CLINICAL TRIAL: NCT06800651
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JMKX003142 in Participants With Rapidly Progressive Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Trial of JMKX003142 in Participants With Rapidly Progressive Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMKX003142-A203
Record Dates: First submitted 2025-01-20; First posted 2025-01-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: ADPKD (Autosomal Dominant Polycystic Kidney Disease)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMKX003142 (Experimental)
  Interventions: Drug: JMKX003142 will be administered orally
- placebo (Placebo Comparator)
  Interventions: Drug: Plcacebo

INTERVENTIONS:
Drug: JMKX003142 will be administered orally — JMKX003142 will be administered orally
  Arms: JMKX003142
Drug: Plcacebo — matched to JMKX003142
  Arms: placebo

SUMMARY:
A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JMKX003142 in Participants with Rapidly Progressive Autosomal Dominant Polycystic Kidney Disease (ADPKD)

DETAILED DESCRIPTION:
Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JMKX003142 in Participants with Rapidly Progressive ADPKD

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the procedures of this trial and provide written informed consent voluntarily;
* Age between 18 to 55 years, male or female;
* ADPKD diagnostic criteria were met before randomization;
* Rapidly progressive ADPKD criteria were met.

Exclusion Criteria:

* 12 weeks prior to screening, patients had taken tolvaptan or another ADPKD improvers, or patients who were assessed by the investigator to be likely to use diuretic during the trial period;
* Praticipants who are unable to feel thirst, or have difficulty with fluid/food intake;
* Patients who have previously received decompression surgery for renal cysts; or who received major surgery within 12 weeks before signing the ICF;
* The investigator think that the praticipant is unable to comply with the requirements of the trial or cannot be evaluated by the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Change of TKV from baseline to Week 52 | 52 weeks

SECONDARY OUTCOMES:
Annual rate of change in eGFR from baseline to Week 52 | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Ph.D, Study Chair — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No